CLINICAL TRIAL: NCT06171997
Title: The Effect of Safe Swaddling After Bathing on Stress and Comfort in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Funda Kardas Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Funda Kardas Ozdemir, Associate Professor, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Funda1
Record Dates: First submitted 2023-11-24; First posted 2023-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2023-12

CONDITIONS: Stress; Comfort
Keywords: Newborn; Bath; Swaddling; Stress; Comfort

STUDY DESIGN:
Intervention Model Description: 36 baby in experimental group and 36 baby in control group, a total of 72 bany will be included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swaddling after bath group (Experimental): Newborns in this group will be swaddled safely after bath.
  Interventions: Other: Swaddling after bath group
- No swaddling after bath group (No Intervention): No action will be taken after bath.

INTERVENTIONS:
Other: Swaddling after bath group — The babies were bathed in the bathtub. Then swaddling was done. The baby was taken into the incubator and waited for 15 minutes. At the end of 15 minutes, the swaddle was opened quietly and slowly, without disturbing the body posture. Stress and comfort scores were given by two observers by video recording the babies before bathing, before swaddling and after swaddling.
  Newborns' stress will be assessed with the Newborn Stress Scale and their comfort with the Newborn Comfort Behavior Scale.
  Arms: Swaddling after bath group

SUMMARY:
The research will be conducted experimentally in the form of randomized controlled studies to determine the effect of safe swaddling of newborns after bathing on stress and comfort. The population of the research consists of newborns receiving treatment and care in the Neonatal Intensive Care Unit of a State Hospital located in the north of Turkey, and the sample consists of 72 babies who meet the sample selection criteria. Descriptive Characteristics Form, Newborn Stress Scale and Newborn Comfort Behavior Scale were used to collect data. Babies will be bathed in the bathtub and then swaddled. The baby will be placed in the incubator and kept for 15 minutes. After 15 minutes, the swaddle will be opened quietly and slowly, without disturbing the body posture. Stress and comfort scores will be given by two observers by video recording the babies before bathing, before swaddling and after swaddling.

DETAILED DESCRIPTION:
Baby bathing is a nursing intervention with individual benefits. Today, there are ongoing discussions about when the infant bath, which is an important part of skin care, should be done first. However, the World Health Organization recommends not bathing newborns for the first 24 hours and waiting until vital signs stabilized. Postponing the bathing of newborns to 48 hours after birth is both effective in maintaining the baby's body temperature and improves skin integrity. Since the thermoregulation abilities of newborns are very limited, it is necessary to maintain body temperature, provide appropriate environmental conditions and warming after bathing.

Although the bathing process, which is an important part of hospital care, protects the health of the newborn, it is also a stressful action for babies and stress symptoms are observed in these babies after bathing. Swaddling the baby in stressful situations such as bathing contributes to the baby's self-calming. The swaddling technique mimics the uterus for newborns and is a technique that ensures the continuation of the intrauterine environment.

Neonatal nursing has come to the forefront in recent years with the development of strategies that increase comfort and has become a frequently used concept in neonatal intensive care units.Among the interventions frequently applied by pediatric nurses to increase comfort are practices such as relaxing positioning, massage, bathing, and wrapping.The practices of nurses to increase the comfort level of the baby and reduce stress with practices with increased level of evidence are very important in terms of nursing care and physical and neuromotor development of the bab.In the light of all this information, this study was planned to investigate the effect of safe swaddling after bathing on stress and comfort in newborns.

ELIGIBILITY:
Inclusion Criteria:

* The week of gestation is between 37 and 41 weeks,
* Birth weight being 2500 g and above,
* Having spontaneous breathing,
* Its physiological parameters are stable,
* Having completed the first 24 hours of life,
* No invasive interventions should be made before the bathing process.

Exclusion Criteria:

Preterms with a gestational age of 22-37 weeks,

* Connected to mechanical ventilator,
* Those who have been wiped or bathed in the last 12 hours,
* Within the first 78 hours of the post-operative period,
* With central catheter,
* Diagnosed with sepsis,
* Those who use sedative and/or muscle relaxants,
* Those with congenital, chromosomal anomalies,

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
change in stress | 15th minute after the procedure
  The Newborn Stress scale will be used to evaluate stress in babies. The scale consists of 8 subgroups including facial expression, body color, respiration, activity level, consolability, muscle tone, extremities and posture, and a total of 24 items in a 3-point Likert type. In scoring, each subgroup is evaluated between 0-2 points. The minimum score obtained from the scale is 0 points and the maximum is 16 points. An increase in the score indicates that the baby's stress level has increased. A change in stress is expected through safe swaddling after bathing compared to before bathing.
change in comfort | 15th minute after the procedure
  Newborn Comfort Behavior Scale (COMFORTneo) will be used to evaluate comfort in babies. It has been stated that the lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6 and the highest score is 30. High scores indicate that the baby is not comfortable and needs interventions to provide comfort. A change in comfort is expected after bathing compared to before bathing through safe swaddling.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Sevgi, RN, Principal Investigator — Kafkas University; Funda Kardaş Özdemir, PhD, Study Director — Kafkas University
Locations (1):
- Kafkas University, Kars, Kars, Turkey (Türkiye)